CLINICAL TRIAL: NCT07058298
Title: An Early Exploratory Clinical Study of GC012F Injection in the Treatment of Refractory Generalized Myasthenia Gravis
Brief Title: GC012F Injection in the Treatment of Refractory Generalized Myasthenia Gravis(24103)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daishi Tian (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Daishi Tian, Chief Physician of Neurology, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC012FinGMG
Record Dates: First submitted 2025-06-07; First posted 2025-07-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Generalized Myasthenia Gravis (gMG)
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3×10^5/kg (Experimental): In this study, the infusion dose of CAR-T cells was set up in one dose group: 3×10^5/kg. About 6 participants are planned to be included. The subjects will be monitored for DLT for 28 days after the infusion of GC012F injection. For the first 3 patients to receive GC012F infusion, if ≤1/3 of the patients develop a DLT at a given dose level, the additional 3 patients will be enrolled in this cohort. If 2/3 or more DLTs occur at this dose level, subsequent subjects may be given a backup dose group of 2.0×10^5/kg or 1.0×10^5/kg after discussion between the investigator and the collaborator.
  Interventions: Drug: GC012F injection

INTERVENTIONS:
Drug: GC012F injection — Subjects will be infused with GC012F Injection within 48-72 hours after lymphodepletion pretreatment,the infusion doses will be (CAR-T cell count) 3 × 10^5/kg.
  Note: for subjects weighing ≤70 kg: number of infused CAR-T cells = 3 (±20%) × 10^5 × body weight(kg); for subjects weighing >70 kg: number of infused CART cells (fixed doses of GC012F Injection) = 3 (±20%) × 10^5 × 70 kg.

SUMMARY:
This is a single-arm, open-label and early exploratory clinical study, with the purpose to study the safety, tolerability and initial clinical efficacy of GC012F Injection in the treatment of refractory GMG and to evaluate the PK, PD characteristics and immunogenicity in subjects with refractory GMG infused with GC012F Injection.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, early-stage exploratory clinical study designed to evaluate safety, tolerability and preliminary efficacy of GC012F injection in the treatment of subjects with refractory GMG,the PK, PD characteristics and immunogenicity of GC012F injection in subjects were evaluated.

This trial is divided into:screening period, apheresis day, baseline period, lymphodepletion pretreatment period, infusion day, safety and efficacy follow-up period, long-term follow-up period and withdrawal visits.Eligible subjects will undergo apheresis collection and then receive the CAR-T infusion after the manufacturing of the products. Subjects in the lymphodepletion cohort will receive the conditioning regimen and then receive CAR-T cell infusion (per the schedule of assessment). Subjects who meet the cell infusion criteria will receive CAR-T cell infusion at the doses levels which were specified in the protocol, and the dose levels could be adjusted according to safety and clinical efficacy.

In this study, the infusion dose of CAR-T cells was set up in one dose group: 3×10^5/kg. About 6 participants are planned to be included. The subjects will be monitored for DLT for 28 days after the infusion of GC012F injection. For the first 3 patients to receive GC012F infusion, if ≤1/3 of the patients develop a DLT at a given dose level, the additional 3 patients will be enrolled in this cohort. If 2/3 or more DLTs occur at this dose level, subsequent subjects may be given a backup dose group of 2.0×10^5/kg or 1.0×10^5/kg after discussion between the investigator and the collaborator.

In the completion dose group of all subjects ,after the DLT observation period, DLTs will be observed for this dose group , all clinical study data collected during the period, especially safety data, were evaluated by the investigator discuss with the collaborator whether to add new subjects to the dose group or explore higher doses group.

After CAR-T cell infusion, subjects will be followed up for safety, cell proliferation, survival, and efficacy until the subject progresses on the disease, or withdraws from the study and refuses to accept follow-up , or dies, or withdraws informed consent, or is lost to follow-up (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled, subjects must meet all of the following criteria:

  1. Subjects or their legal representatives voluntarily sign a written informed consent and are willing and able to comply with the procedures of the study;
  2. Subjects aged 18-75 years old (both inclusive), male or female;
  3. Subjects with confirmed refractory gMG of classes IIa - IVb by MGFA clinical classification (including classes IIa, IIb, IIIa, IIIb, IVa and IVb) at screening;
  4. Subjects with the Myasthenia Gravis - Activities of Daily Living (MG-ADL) score of ≥6, the proportion of ocular symptoms of <50% of the total score, and the Quantitative Myasthenia Gravis (QMG) score of ≥11;
  5. Subjects with poor response and/or who do not respond to the conventional therapies, that means subjects who are still at risk of relapse or exacerbation after conventional therapies with hormones, immunosuppressants (e.g., azathioprine, mycophenolate mofetil, tacrolimus, cyclosporin A, cyclophosphamide, methotrexate, etc.), or biological agents (e.g., rituximab);
  6. For patients who are taking corticosteroids, the dose of prednisone should not exceed 30 mg/day (or an equivalent dose of other corticosteroids), and the dose must be stable for at least 4 weeks before infusion;
  7. The laboratory test results during the screening period meet the following criteria:

     1. Neutrophil count ≥ 1.0×10^9/L; Hemoglobin ≥ 8.0 g/dL; Platelet count≥50×10^9/L;
     2. Alanine aminotransferase ≤ 3× upper limit of normal (ULN); Aspartate aminotransferase ≤ 3×ULN; total bilirubin (TBIL) < 2× ULN (for subjects with Gilbert's syndrome), direct bilirubin (DBIL)) ≤ 1.5×ULN
     3. Creatinine clearance (19.3 Appendix 3) ≥ 30 mL/min;
     4. Activated partial thromboplastin time (APTT) ≤ 1.5×ULN, prothrombin time (PT)≤ 1.5×ULN;
     5. Subject's left ventricular ejection fraction (LVEF) is ≥ 50% by echocardiography, with no evidence of pericardial effusion as determined;
  8. Female subjects of child-bearing age must:

     1. At screening, a negative serum β human chorionic gonadotropin β-hCG pregnancy test result confirmed by the investigator;
     2. Who agree to avoid breastfeeding during the study period until at least 1 year after the infusion of GC012F Injection or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later).
  9. Male subjects with sexual partners and female subjects of potential child-bearing age shall agree to take effective contraceptive measures (e.g., oral contraceptive pills, intrauterine device or condom) from the screening period until at least 2 years after the infusion of GC012F Injection or until two consecutive flow cytometry tests show the absence of CAR-T cells (whichever occurs later). Male subjects must agree to use condoms during sexual contact with pregnant women or females of child-bearing age within at least 2 years after the infusion of GC012F Injection, even if a successful vasectomy has been performed;
  10. Subjects for whom venous access available for blood collection can be established, and with no contraindications to leukocyte collection.

Exclusion Criteria:

* Participants who meet any of the following criteria are not included in the study:

  1. Have a history of severe hypersensitivity or allergy;
  2. Contraindications or hypersensitivity to fludarabine, cyclophosphamide and any component of the test drug;
  3. Subjects who have received intravenous immunoglobulin or plasma exchange therapy or immunoadsorption therapy within 4 weeks prior to infusion;
  4. Received CD20-targeted drugs within 6 months prior to apheresis;
  5. Received Tacrolimus, Cyclosporine, Azathioprine, Mycophenol Mofetil within 1 week before apheresis;
  6. Treatment with neonatal Fc receptor (FcRn) antagonists within 1 week prior to apheresis;
  7. Patients who have received complement inhibitors (e.g., eculizumab, etc.) within 1 weeks before apheresis ;
  8. Subjects with any of the following heart diseases:

     1. Class III or Class IV congestive heart failure based on New York Heart Association (NYHA) Functional Classification;
     2. Unstable angina, myocardial infarction or coronary artery bypass grafting (CABG) within 6 months prior to screening;
     3. Clinically significant ventricular arrhythmia or a history of unexplained syncope not due to vasovagal reaction or dehydration; or a QTc interval >480 ms at screening;
     4. Has a history of severe non-ischemic cardiomyopathy;
     5. Severe cardiovascular abnormalities (such as brain natriuretic peptide (BNP)/troponin and other indices) and the investigator judges that such subjects are not eligible for enrollment.
  9. Subjects with other uncontrolled malignancies. The following conditions will be excluded: early-stage tumors that have been treated by radical surgery (carcinoma in situ or grade 1 tumors, or non-ulcerative primary melanoma with a depth of <1 mm and with no involvement of lymph nodes), basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in situ, or breast cancer in situ that has been treated by potential radical treatment;
  10. Serious underlying medical conditions, such as:

      1. Viral, bacterial, fungal, or other infections that are uncontrollable or requiring systemic intravenous therapy (including tuberculosis infection with clear evidence of disease activity) as demonstrated by evidence;
      2. Dementia or mental status changes as demonstrated by significant clinical evidence;
      3. History of any central nervous system (CNS) or neurodegenerative diseases, (e.g., Epilepsy, Convulsion, Paralysis, Aphasia, Stroke, Severe brain injury, Dementia, Parkinson's disease, Mental Illness).
  11. Positive result for any of the following tests:

      1. Positive test result of human immunodeficiency virus (HIV) antibody;
      2. Positive test result of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) (HBV DNA copy number will be detected for HBcAb- or HBsAb-positive patients. If the copy number is lower than the lower limit of detection, patients can be enrolled under the premise of standardized antiviral therapy);
      3. Positive test result of hepatitis C virus (HCV) antibody with the copy number of HCV RNA higher than the lower limit of detection; or with known history of hepatitis C without completion of antiviral therapy for ≥24 weeks;
      4. Positive test result of Syphilis antibody.
  12. Prior treatment with a CAR-T product for any target;
  13. Previous organ or allogeneic bone marrow transplantation;
  14. Subjects who have undergone surgery within 2 weeks prior to lymphodepletion pretreatment or plan to undergo surgery during the study (except subjects who schedule for local anesthesia surgery, but the surgery cannot be performed within 2 weeks after infusion);
  15. Received live attenuated vaccine within 4 weeks prior to lymphodepletion pretreatment;
  16. Subjects who have received study drugs in other clinical trials within 4 weeks prior to signing the informed consent form, or whose ICF signing date is within 5 half-lives of the last dose they had taken in other clinical trial (whichever is longer);
  17. Pregnant females or lactating females who do not agree to give up breastfeeding, during the period of participation in this study or men with a family plan within 1 year of receiving study treatment and females;
  18. Subjects with suicidal intentions at present based on the Columbia-Suicide Severity Rating Scale (C-SSRS), i.e., the answer to Question 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on "Suicide" in the C-SSRS is "Yes", or who have a history of suicidal behavior at present;
  19. According to the researcher's judgment, there are circumstances that may prevent the subject from participating in the full trial, confuse the trial results, or participation in this study is not in the best interests of subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-02-13 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of adverse events. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.

SECONDARY OUTCOMES:
Analysis of cell dynamics (CK) parameters of the copy number of the GC012F CAR gene in peripheral blood- Cmax(based on data availability). | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Analysis of cell dynamics (CK) parameters of the copy number of the GC012F CAR gene in peripheral blood- Tmax(based on data availability). | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Analysis of cell dynamics (CK) parameters of the copy number of the GC012F CAR gene in peripheral blood- AUC(based on data availability). | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
T/B lymphocyte subsets in peripheral blood after GC012F infusion. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Levels of cytokines in peripheral blood after GC012F infusion. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Proportion of patients with improvement in MG-Activities of Daily Living (MG-ADL) score and quantitative muscle weakness (QMG) score and MG-ADL and QMG score with different improvement scores from baseline to 24 weeks after GC012F infusion. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Proportion of patients with MG composite score (MGC) improvement and MGC score improvement scores from baseline to 24 weeks after infusion and reinfusion of GC012F. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Mean change in patient-reported outcome scores such as MG-QoL15r score from baseline to 24 weeks after infusion and return infusion of GC012F. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Change in the patient's status after MGFA intervention 24 weeks after the infusion of GC012F. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
Reduction in pathogenic antibody levels and proportion of patients in a cohort of MG-specific autoantibody-positive patients from baseline to 24 weeks after GC012F infusion and reinfusion. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.

OTHER OUTCOMES:
To evaluate the immunogenicity of GC012F injection | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
  The changes in serum immunoglobulin concentrations (including IgG, IgM, IgA, and IgE) within 24 weeks after the infusion of GC012F.
To evaluate immune reconstitution after infusion of GC012F injection | Since signing the ICF until 24-week post-infusion or premature withdrawal from the study, whichever comes first.
  Incidence and titer of anti-CAR AZD0120 antibody response during the study period.
To determine the presence of replication competent lentivirus (RCL) and lentiviral integration site in subjects after infusion of GC012F lnjection. | Since signing the ICF until 24-week post-infusion or withdrawal from the study, whichever comes first.
  Detection rate of RCL

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical Colledge, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No